CLINICAL TRIAL: NCT06165289
Title: Efficacy and Safety of Endoscopic Balloon Dilatation Combined With Autologous Platelet-rich Plasma (PRP) Injection in Colonic Stenosis in Crohn's Disease
Brief Title: Endoscopic Balloon Dilatation Combined With PRP Injection in Colonic Stenosis in Crohn's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: luyi45
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP high concentration group (Experimental): Endoscopic balloon dilatation combined with autologous platelet-rich plasma (PRP) injection with high concentration (platlet 2*10^6/μL)
  Interventions: Other: PRP Injection
- PRP low concentration group (Experimental): Endoscopic balloon dilatation combined with autologous platelet-rich plasma (PRP) injection with low concentration (platlet 1*10^6/μL)
  Interventions: Other: PRP Injection

INTERVENTIONS:
Other: PRP Injection — Endoscopic balloon dilatation combined with autologous platelet-rich plasma (PRP) injection with different concerntrations

SUMMARY:
The aim was to investigate whether endoscopic balloon dilatation combined with PRP injection can help prevent or prolong restenosis in patients with Crohn's disease with colonic stenosis, and to explore the concentration of PRP. The study was a single-center, randomized, non-controlled study. Experimental group of patients underwent endoscopic balloon dilation and submucosal injection of PRP at the wound edge, historical control was used, and the patients included in the study were randomly divided into high concentration group and low concentration group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as CD;

  * Stenosis of the colon was found during colonoscopy, and surgery was not considered for the time being; ③ Narrow length <5cm; ④ The patients agreed to undergo endoscopic balloon dilatation and voluntarily signed the informed consent to participate in this study, and were capable of complying with the agreement.

Exclusion Criteria:

* The patient has contraindications for endoscopic therapy, such as coagulation disorder, severe cardiopulmonary dysfunction, active bleeding, and inability to cooperate.

  * Deep and large active ulcer was found in the stenosis;

    * < 18 years old;

      * Foreign patients;

        * Patients with a history of malignant tumors, including melanoma (except local skin cancer);

          * Pregnant or nursing patients;

            * Patients who could not be followed at all nodes of the primary outcome indicator; Other diseases that researchers believe could put patients at risk;

              * Other diseases that researchers believe could put patients at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
restenosis rate | 3 months after endotherapy
  restenosis means the endoscopy with size of 10.5mm can not pass the stricture afer endotherapy

SECONDARY OUTCOMES:
Changes in intestinal ultrasound | 3 months after endotherapy
  the thickness of the stricture intestinal wall, and the width of the proximal intestinal cavity
Proportion of surgery | 1 year after endotherapy
  The proportion of surgery due to stenosis or perforation

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No